CLINICAL TRIAL: NCT05817617
Title: Vitamin D and Head and Neck Cancer: Impact on Toxicity and Prognosis: Prospective Multicenter Study of Head-Neck Group of the Italian Association of Radiotherapy and Clinical Oncology (AIRO)
Brief Title: Vitamin D and Head and Neck Cancer: Impact on Toxicity and Prognosis
Status: Recruiting | Type: Observational
Sponsor: Centro di Riferimento Oncologico - Aviano (Other)
Responsible Party: Sponsor
Other Study IDs: CRO 2021.013
Record Dates: First submitted 2023-03-24; First posted 2023-04-18 (Actual); Last update posted 2023-10-25 (Actual); Status verified 2023-04

CONDITIONS: Head and Neck Cancer
MeSH Terms: conditions — Head and Neck Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Head and Neck cancer patients: candidate to receive definitive or adjuvant radiation therapy with bilateral neck irradiation

SUMMARY:
The goal of this observational study is to learn about relation between vitamin D levels in subjects with head and neck cancer. The main question it aims to answer are:

* variation of vitamin D levels in the study population at different time points
* relation between therapy side effects and vitamin D level
* relation between disease outcome and vitamin D level Participants will be followed as per clinical practice

DETAILED DESCRIPTION:
There are only a few works in the literature that correlate the circulating levels of vitamin D with the prognosis or development of toxicity in treated HNSCC patients with radical intent radiation therapy. These small studies have highlighted a worse outcome and greater toxicity in patients with low vitamin D levels. The study aims to study the variations in circulating levels of vitamin D in a multicenter cohort of patients with HSNCC prospectively collected and to evaluate the impact of vitamin D levels at diagnosis on the development of toxicity and on disease outcome

ELIGIBILITY:
Inclusion Criteria:

histologically proven HNSCC (squamous cell carcinomas), all subsites

* non-metastatic locally advanced stages
* patients candidate for radical or adjuvant radiotherapy
* patients candidate for bilateral neck irradiation
* written informed consent

Exclusion Criteria:

* distant metastases
* patients with known disorders of calcium/vitamin D metabolism

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients of the participant centers with histologically proven HNSCC (squamous cell carcinomas)
Sampling Method: Non-Probability Sample
Enrollment: 953 (Estimated)
Dates: Start 2021-08-08 (Actual); Primary Completion 2024-08 (Estimated); Study Completion 2026-08 (Estimated)

PRIMARY OUTCOMES:
Vitamin D variation | 7 weeks
  Difference in vitamin D levels between baseline and during radiotherapy

SECONDARY OUTCOMES:
Baseline vitamin D level and radiotherapy toxicity | 8 weeks
  Evaluation of the impact of baseline vitamin D levels on acute toxicity (mucositis, dermatitis and weight loss >10%)
Baseline vitamin D level and response | 12 weeks
  Evaluation of the impact of baseline vitamin D levels on response measured in term of ORR (Objective Response Rate)
Baseline vitamin D level and relapse free survival | up to 2 years
  Impact of baseline vitamin D levels on relapse free survival
Baseline vitamin D level and survival | up to 2 years
  Impact of baseline vitamin D levels on overall survival
Variation of vitamin D level | 4 weeks
  Difference and relation between vitamin D levels at baseline and after 4 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Giuseppe Fanetti, MD, Principal Investigator — Centro di Riferimento Oncologico (CRO), IRCCS
Locations (10):
- Italy (10):
  - Ospedale Mons AR Dimiccoli, Barletta, BAT
  - Centro di Riferimento Oncologico - Aviano, Aviano, Pordenone
  - Ospedale dell'Angelo, Mestre, Venezia
  - Ospedali Riuniti, Ancona
  - AORN San Pio, Benevento
  - IEO, Milan
  - Ospedale Niguarda, Milan
  - Ospedale del Mare, Napoli
  - Azienda Ospedaliero Universitaria di Pisa, Pisa
  - Policlinico Umberto I, Roma

IPD SHARING:
Plan to Share IPD: No
No sharing